CLINICAL TRIAL: NCT00270088
Title: A Double-Blind, Placebo-Controlled Study to Determine Whether Procrit� (Epoetin Alfa) Can Reduce Peri-Operative Transfusion Requirements in Subjects Undergoing Major Orthopedic Surgery
Brief Title: A Study to Determine Whether Epoetin Alfa Can Reduce the Need for Blood Transfusions in Patients During the Period of Time Around Major Orthopedic Surgery.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR005899
Record Dates: First submitted 2005-12-22; First posted 2005-12-26 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2011-02

CONDITIONS: Anemia; Blood Transfusion; Orthopedic Procedures
Keywords: Anemia; blood transfusion; epoetin alfa; epogen; erythropoietin; orthopedic procedures; orthopedic surgery
MeSH Terms: conditions — Anemia | interventions — Epoetin Alfa

INTERVENTIONS:
Drug: epoetin alfa

SUMMARY:
The purpose of this study is to evaluate the safety of epoetin alfa and to determine whether epoetin alfa will reduce the need for blood transfusions during the period of time around major orthopedic surgery. Epoetin alfa is a genetically engineered protein that stimulates red blood cell production.

DETAILED DESCRIPTION:
Patients undergoing major orthopedic surgery frequently require blood transfusions both during and after the operation. These transfusions can result in adverse reactions, such as a blood clot in a deep vein. Agents that can reduce the need for transfusions would improve the overall safety of the surgery. In previous studies with epoetin alfa, patients have generally experienced an increase in the percentage of red blood cells in whole blood, a decrease in blood transfusions, and a decrease in the number of surgery-related adverse reactions, with good tolerance of the drug. This is a randomized, double-blind, placebo-controlled, parallel group, multicenter study. The study will evaluate the safety of epoetin alfa and to determine whether epoetin alfa will reduce the need for blood transfusions in patients who are expected to require at least 2 units of blood during the period of time around major orthopedic hip or knee surgery. Before the start of the study, patients are screened for eligibility and a test is performed to determine the amount of hemoglobin present in each patient's blood. Based on these results, patients are then divided into 3 groups: patients with hemoglobin <=10 grams/deciliter (g/dL), patients with hemoglobin >10 and <=13 g/dL, and patients with hemoglobin >10 g/dL. Within each of these groups, patients will be randomly assigned to receive 1 of 3 treatments: epoetin alfa 300 units/kilogram (U/kg), epoetin alfa 100 U/kg, or placebo, by injection beneath the skin, beginning 10 days before scheduled surgery and ending 4 days after surgery. Additionally, from 10 days before surgery until 4 days after surgery all patients will receive a 150 milligram iron supplement daily by mouth, and from the day of surgery (following surgery) until 6 days after surgery, all patients will be given Coumadin 5 milligrams daily (a drug to prevent a blood clot in a deep vein). Safety evaluations include laboratory tests, physical examination, vital signs, and the recording of adverse events performed throughout the study until the patient is discharged from the hospital. In addition, six weeks after surgery, laboratory tests are performed, vital signs are measured, and any adverse events are recorded. Ultrasound is performed before the start of the study and on Day 5 after surgery to determine if there is a blood clot in a deep vein. Effectiveness will be determined by reduction in the need for transfusions during the period of time around the surgery. The study hypothesis is that patients treated with epoetin alfa will require fewer transfusions during the period of time around surgery than patients treated with placebo. Epoetin alfa 300 units/kilogram (U/kg), epoetin alfa 100 U/kg, or placebo, by injection beneath the skin beginning 10 days before scheduled surgery and ending 4 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for major orthopedic surgery involving the hip or knee, who are expected to require transfusion of at least 2 units of red blood cells
* who are unwilling or unable to participate in a transfusion program wherein a patient's own blood is donated before surgery
* in good general health
* having no significantly abnormal laboratory blood, urine, or stool tests

Exclusion Criteria:

* Patients having any blood disease, hepatitis B, signs and symptoms suggestive of an autoimmune disease causing blood to break down and release iron-containing pigment, or who have tested positive for HIV (human immunodeficiency virus)
* who are unable to use Coumadin (a medication to prevent blood clots in veins)
* having a recent history of stomach or intestinal bleeding, bleeding inside the skull, or the signs and symptoms of significant and ongoing blood loss
* having a seizure disorder, uncontrolled high blood pressure, the presence of active inflammatory disease (i.e., rheumatoid arthritis, however, patients with osteoarthritis may be included in this study) or the signs and symptoms of a significant disease and/or dysfunction
* received a blood transfusion within 1 month before the start of the study, received medication known to suppress formation of red blood cells within 1 month before the start of the study, or having infections or cancers that may make it difficult to respond to the study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Actual)
Dates: Start 1993-04; Study Completion 1994-08 (Actual)

PRIMARY OUTCOMES:
Proportion of patients in each treatment group, overall, and within each baseline hemoglobin group requiring blood transfusion following major orthopedic surgery

SECONDARY OUTCOMES:
Changes in hemoglobin, hematocrit, and red blood cell count; Assessment of safety (laboratory tests, vital signs, and physical examination from start to end of study); Assessment of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A study to determine whether epoetin alfa can reduce the need for blood transfusion in patients during the period of time around major orthopedic surgery — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=679&filename=CR005899_CSR.pdf